CLINICAL TRIAL: NCT02366780
Title: Breast Milk Content Expressed Manually Compared to Electric Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SD-0662-11-TLV
Record Dates: First submitted 2015-02-04; First posted 2015-02-19 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Infant
Keywords: Lactation; Breastmilk; Macronutrients
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual expression followed by electric pump (Experimental): Mothers will be assigned to first express breast milk manually followed by electric pump
  Interventions: Procedure: Pump
- Electric pump followed by manual expression (Experimental): Mothers will be assigned to first express breast milk by electric pump followed by manual expression
  Interventions: Procedure: Pump

INTERVENTIONS:
Procedure: Pump — Breast milk expression using manually or using an electric pump

SUMMARY:
Breast milk is a unique and unmatched nutritional and non-nutritive source of bioactive factors for the health and development of infants.Colostrum, which is produced in low quantities for the first 3 to 4 days after birth, is rich in immunologic components and developmental factors.

Breastfeeding difficulties during the first days of life of an infant are common. Moreover, not all infants can be directly fed at the breast.

Therefore, breast milk feeding at this early stage is initiated and promoted by the expression of breast milk either manually or by use of a pump. Whether the method of milk expression at this stage has a qualitative impact on colostrum is currently unknown.

The purpose of this randomized controlled study is to compare the effect of manual expression with electric pump expression upon the macronutrient composition of breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy lactating mothers of term infants

Exclusion Criteria:

* HIV infected mothers

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Macronutrient content of expressed breast milk | 3 to 5 min
  Mothers will express milk from the same breast indicated in the assigned arm. Macronutrient content will be analyzed using the Human Milk Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Dolberg, MD, Principal Investigator — Department of Pediatrics, Sakler Faculty of Medicine
Locations (1):
- Department of Neonatology, Lis Maternity Hospital, Tel Aviv medical Center, Tel Aviv, Israel

REFERENCES:
- [Result] Mangel L, Ovental A, Batscha N, Arnon M, Yarkoni I, Dollberg S. Higher Fat Content in Breastmilk Expressed Manually: A Randomized Trial. Breastfeed Med. 2015 Sep;10(7):352-4. doi: 10.1089/bfm.2015.0058. Epub 2015 Jul 14. PMID 26171639